CLINICAL TRIAL: NCT05142358
Title: A Prospective Study to Evaluate Continuous Positive Airway Pressure Devices to Reduce Pulmonary Dose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5Y21
Record Dates: First submitted 2021-10-04; First posted 2021-12-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Left Sided Breast Cancer
Keywords: stereotactic body radiation therapy; continuous positive airway pressure; CPAP; radiation; cancer; lung; Deep inspiratory breath hold (DIBH)
MeSH Terms: conditions — Lung Neoplasms; Unilateral Breast Neoplasms; Neoplasms | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: All participants will undergo standard of care radiation treatment. One additional CT scan will be performed with the use of a CPAP device to determine effect on dosimetry.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- left-sided breast cancer (Active Comparator): Participants will come in for their regularly scheduled radiation planning and treatment. Participants will undergo three scans (with and without DIBH (i.e., free-breathing), with CPAP). Participants will also use the CPAP device before the CT scan, for which they will be educated and trained.
  Interventions: Device: Continuous Positive Airway Pressure; Other: Deep inspiratory breath hold; Other: Free Breath
- Lung SBRT (Active Comparator): Participants will come in for their regularly scheduled radiation planning and treatment. Participants will undergo three scans (with and without DIBH (i.e., free-breathing), with CPAP). Participants will also use the CPAP device before the CT scan, for which they will be educated and trained.
  Interventions: Device: Continuous Positive Airway Pressure; Other: Deep inspiratory breath hold; Other: Free Breath

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Use of CPAP device at the start of treatment planning.
  Other Names: CPAP
Other: Deep inspiratory breath hold — Treatment during breath holds leads to longer treatment times for patients and radiation oncology departments
  Other Names: DIBH
Other: Free Breath — Regular breathing
  Other Names: Without DIBH

SUMMARY:
Data collection and assessment on patients with left-sided breast cancer or undergoing lung stereotactic body radiation therapy (SBRT) utilizing continuous positive airway pressure (CPAP) devices.

DETAILED DESCRIPTION:
Lung stereotactic body radiation therapy (SBRT) has emerged as a definitive treatment for patients with early-stage lung cancers as well as for patients with limited metastases to the lung. One challenge with the treatment of the lung is the risk of pulmonary toxicity, particularly for early-stage lungs cancers that are inoperable (those receiving primary lung SBRT) or those with metastatic cancers receiving systemic therapy that may impact pulmonary function (those receiving lung SBRT for metastatic cancers).

Continuous positive airway pressure (CPAP) devices are commonly utilized for patients with obstructive sleep apnea. However, through the use of continuous pressure, lung volumes are increased. Preliminary data in patients undergoing breast radiation as well as lung radiation has demonstrated the safety and feasibility of such an approach, demonstrating increased lung volumes with decreases in heart dose6-8. Additional potential advantages of CPAP include increased ease of use for patients and the potential for cost savings as compared to traditional respiratory management techniques.

This prospective study is to allow for the collection and assessment of data on patients with left-sided breast cancer or undergoing lung SBRT utilizing CPAP. This will allow for the assessment of lung doses with and without CPAP as well as cardiac doses. No additional changes to our standard of care breast or lung radiation will occur. With respect to the safety profile, CPAP is commonly used with limited toxicity concerns. The potential benefit of CPAP has reduced lung and heart doses and, consequently, radiation-related toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with left-sided breast cancers

  * Patients must be undergoing left breast/chest wall radiation with or without regional nodal irradiation
* Patients undergoing lung SBRT

  * Primary lung cancers
  * Metastatic lung tumors

Exclusion Criteria:

* Patients with right side breast cancer
* Patients who are unable to tolerate the CPAP device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Dosimetry comparison CPAP and free breathing. | At the time of Scan, " Day 1"
  The primary objective will be to assess changes in lung dosimetry V5 on the affected side when using CPAP compared to free breathing will be measured in percentages.
Dosimetry comparison CPAP and free breathing. | At the time of Scan, " Day 1"
  The primary objective will be to assess changes in lung dosimetry V20 on the affected side when using CPAP compared to free-breathing will be measured in percentages.
Dosimetry comparison CPAP and free breathing. | At the time of Scan, " Day 1"
  The primary objective will be to assess changes in lung dosimetry mean lung on the affected side when using CPAP compared to free-breathing will be measured in Grays.

SECONDARY OUTCOMES:
Total Lung dosimetry | At the time of Scan, " Day 1"
  Total Lung dosimetry will be measured in Grays.
Cardiac dosimetry with CPAP as compared to free breathing | At the time of Scan, " Day 1"
  Cardiac dosimetry with CPAP as compared to free-breathing will be measured in Grays.
Measure breast/chest wall or lung tumor motion as well as organ at risk motion | At the time of Scan, " Day 1"
  Simulation scans will be performed with CPAP and free breathing. The breast/chest wall, and tumors (lung SBRT), as well as lung and heart, will be contoured on each scan. Using the CPAP scan as a reference, we will assess breast/chest wall motion, lung tumor motion, and organ at risk (ex. heart, abdominal organs) motion with free-breathing scans for each patient and analyze by treatment site (breast vs. lung SBRT).
Treatment time with CPAP treatments | At the time of Scan, " Day 1"
  Treatment time will be measured for each fraction
Confirm maintenance of inflation with CPAP using surface guidance | At the time of Scan, " Day 1"
  At the time of simulation, investigators will create a surface rendering with the patient using CPAP. Investigators will assess maintenance of inflation when using CPAP where all three dimensions will be measured during treatment by comparing the surface rendering obtained during simulation with CPAP to the surface during treatment with CPAP, assessing for the greatest changes over the course of each fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Sheeh Cherian, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States